CLINICAL TRIAL: NCT05143177
Title: An Adaptive Phase 2/3 Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel, 2 Arm Study to Evaluate the Efficacy and Safety of DA-1229 (Evogliptin) in Patient's Calcific Aortic Valve Disease With Mild to Moderate Aortic Stenosis (EVOID-AS)
Brief Title: A Study to Evaluate the Efficacy and Safety of DA-1229 (Evogliptin) in Patient's Calcific Aortic Valve Disease With Mild to Moderate Aortic Stenosis (EVOID-AS)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: REDNVIA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR-CAVD-001
Record Dates: First submitted 2021-10-20; First posted 2021-12-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Calcific Aortic Valve Disease
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DA-1229 10 mg (Active Comparator)
  Interventions: Drug: Evogliptin

INTERVENTIONS:
Drug: Evogliptin — DA-1229 10 mg, 1 tab
  Other Names: DA-1229
  Arms: DA-1229 10 mg
Drug: Placebo — DA-1229 Placebo, 1 tab
  Arms: Placebo

SUMMARY:
This is an adaptive Phase 2/3 multicenter, double-blind, placebo-controlled, randomized, parallel, 2 arm study to evaluate the efficacy and safety of DA-1229 compared to placebo in patients with calcific aortic valve disease with mild to moderate aortic stenosis. There are 2 arms in this study to which patients will be randomized in a ratio of 1:1 to receive the DA-1229 or placebo orally once daily for a period of 104 weeks. The 2 arms are: placebo and DA-1229 10 mg Group.

The study will have three phases: Screening Period (up to 4 weeks), Treatment Period (104 weeks), and Follow-Up Period (2-4 weeks). Total Study Duration is112 Weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 35 years of age at time of screening.
2. Subject has calcific aortic valve disease with mild to moderate aortic stenosis as defined by

   * Doppler echocardiography results: Aortic Valve mean pressure gradient between 10-30 mmHg and Aortic Valve Area ≥ 1.2 and ≤ 2.0 cm2 on TTE within 2 weeks prior to randomization and,
   * Cardiac Compute Tomography (CT) test results: aortic valve calcium score (AVCS) ≥ 200 AU at baseline cardiac CT within 4 weeks prior to randomization
3. Subject provides written informed consent prior to initiation of any study procedures.
4. Subject understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Subject has concomitant moderate or more aortic valve regurgitation.
2. Subject has concomitant moderate or severe mitral or tricuspid valve disease.
3. Subjects has left ventricular ejection fraction < 50%.
4. Subject previous history of aortic valve surgery.
5. Subject has NYHA class III or IV heart failure.
6. Subjects whose alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal range.
7. Subjects who cannot undergo Cardiac CT.
8. Subjects whose life expectancy is < 2 years.
9. Subjects with ESRD (End-stage Renal Disease) defined as eGFR (calculated using MDRD equation) ≤ 30 mL/min/1.73m2 or in need of dialysis.
10. Subject has Type 1 diabetes mellitus.
11. Subject has a history of diabetic ketoacidosis (DKA).
12. Subject has a history of severe hypoglycemia (blood glucose levels < 54 mg/dl) within the previous six months prior to screening.

    Note: Subjects receiving treatment for their non-type 1 diabetes and without history of DKA or severe hypoglycemia episode in the preceding 6 months who are interested in participating in the trial are recommended to inform/consult their diabetes provider prior to enrollment in the study or IP initiation to discuss if adjustment in their diabetes therapy or other monitoring may be needed.
13. Subject has pancreatic Amylase isoenzyme and/or Lipase elevation ≥ 3x the upper limit of normal (ULN) at screening or baseline visit, or subject has a history of pancreatitis
14. Subjects who are currently taking or anticipated to take any of the following medications for the duration of the study:

    oDPP4 inhibitor other than the investigational product

    ▪Subjects taking insulin or sulfonylureas should consult their primary diabetes provider prior to enrollment in the study or IP initiation to discuss if adjustment in their diabetes therapy and/or other monitoring may be needed.

    oVitamin K

    ▪Subjects taking over-the-counter multivitamins containing ≤ 90 mcg/day vitamin K will be allowed to continue use during the study.

    oChronic use of any medications that strongly impact hepatic metabolism by way of inducing or inhibiting the CYP3A4 system, giving rise to drug-drug interaction (with the exception of focal or limited topical treatment)
    * Strong CYP3A4 inducers* including but not limited to barbiturates (phenobarbital), rifampicin/rifabutin, carbamazepine, phenytoin, primidone, St. John's Wort, Efavirenz, griseofulvin, and chronic (>1 month) supraphysiologic glucocorticoid use (>7.5 mg/day prednisone or equivalent glucocorticoid dosing).
    * Strong CYP3A4 inhibitors*including but not limited to protease inhibitors for treatment of HIV/HCV (such as ritonavir, lopinavir, atazanavir, etc.), chronic systemic use of azole antifungals (ketoconazole, fluconazole, itraconazole, voriconazole) and clarithromycin Note: Short-term/temporary use of clarithromycin, azole antifungals or Paxlovid (for treatment of COVID-19) is allowed, but temporary study drug hold during the course of these treatment would be necessary.
15. Subjects with history of severe allergic reaction to DPP4 inhibitors including anaphylaxis and angioedema.
16. Subjects with galactose intolerance, lapp lactase deficiency, and glucose-galactose malabsorption.
17. Subjects with history of severe cerebrovascular diseases (such as cerebral infarction or transient ischemic attack), severe cardiovascular diseases (such as unstable angina, myocardial infarction and life-threatening arrhythmia) within 6 months of screening.
18. Subjects with history of malignant tumor within the past 3 years prior to Screening Visit (Visit 1) unless cure is expected.
19. Subjects with history of drug or alcohol abuse. History of cannabis/Marijuana use including recreational use in the last 6 months and an unwillingness to abstain during the course of the study.

    oNote: Alcohol abuse is a pattern of drinking that results in harm to one's health, interpersonal relationships, or ability to work. Manifestations of alcohol abuse include the following: Failure to fulfill major responsibilities at work, school, or home, drinking in dangerous situations, such as drinking while driving or operating machinery, legal problems related to alcohol, such as being arrested for drinking while driving or for physically hurting someone while drunk and continued drinking despite ongoing relationship problems that are caused or worsened by drinking
20. Subjects with history of medication non-compliance.
21. Pregnant or lactating women.
22. Subjects who used investigational drugs or devices within 4 weeks or investigational biologics within the last 6 months prior to screening and for the duration of the study.
23. Inability to provide informed consent or to comply with test requirements.
24. Subjects with physical (severe hepatic, cardiac, renal, pulmonary, hematological, endocrine, gastrointestinal, etc. conditions) or mental (cognitive, psychiatric, etc. conditions) conditions that may impact their ability to take part in the study.
25. Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment.
26. Women of child-bearing age who are sexually active but decline to take proper contraceptive measures during the study period, unless the female is post-menopausal for at least 2 years or are surgically sterile.

    * Note: Women of childbearing potential (WOCBP) and Women not of childbearing potential are eligible to participate. Women of childbearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 30 days after taking the last dose of investigational product).
    * Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile or 2 years post-menopausal. All male subjects/partners of WOCBP must agree to consistently and correctly use a condom for the duration of the study and for 30 days after taking the study drug. In addition, subjects may not donate ova or donate sperm for the duration of the study and for 30 days after taking the last dose investigational product.

Withdrawal Criteria:

A subject who is randomized into the study, but who does not complete the study will be considered prematurely discontinued.

At any point during the study all subjects have the right to withdraw without prejudice to future care. Documentation to whether or not each subject completed the clinical study will be recorded. If for any subject, study treatment was discontinued, the reason(s) will be documented.

The Investigator can discontinue a subject at any time if in their clinical judgment it is considered to be medically necessary. Investigators considering discontinuing study treatment should contact the medical monitor prior to such discontinuation. Subjects who have study treatment discontinued will continue to be followed per protocol (i.e., to complete EOT Visit and Visit 11 assessments), whenever possible. Subjects who have study treatment discontinued due to a serious adverse event will be followed until resolution or stabilization of the event. Reasons for subject withdrawal/discontinuation may constitute one of the following:

* Voluntary withdrawal of his/her informed consent
* Administration of any prohibited medication unless otherwise approved by the investigator(s)
* Serious adverse event or adverse drug reaction that causes withdrawal from the study, such as development of acute pancreatitis investigator(s)
* Any evidence of pancreatic inflammation on pancreatic imaging (CT Scan or Magnetic resonance cholangiopancreatography (MRCP) or Ultrasound)
* Severe breach against this protocol such as breach of any inclusion or exclusion criteria
* When Investigator judges aortic valve surgery or procedure is necessary due to progression of disease as per the Critical Pathways presented in American and European Society of Cardiology
* Failure to trace the subject - out of contact, etc. - for follow-up observation
* Pregnancy
* Discontinuation of study by the Sponsor

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Aortic valve calcification as measured by change from baseline in Agatston arbitrary unit (AU) using cardiac computed tomography (CT) at 104 weeks | at 104 weeks

SECONDARY OUTCOMES:
Change in aortic stenosis severity as measured by mean pressure gradient using echocardiography at week104 as compared to baseline | at week104
Change in aortic stenosis severity as measured by aortic valve area (AVA) using echocardiography at week 104 as compared to baseline | at week104
Time-to-AV intervention to treat aortic stenosis including AV replacement | at week104

OTHER OUTCOMES:
Time-to-major adverse cardiovascular events of cardiac death, non- fatal myocardial infarction, heart failure hospitalization and stroke | at week 104 as compared to baseline
Time-to-symptom onset | at week 104
Aortic valve calcification as measured by change from baseline change from baseline in Arbitrary Units (-AU) by the Agatston method using cardiac computed tomography (CT) at week 52 | at week 52
Change in aortic stenosis severity as measured by aortic valve area (AVA) using echocardiography at week 52 as compared to baseline | at week 52
Change in aortic stenosis severity as measured by peak transaortic velocity using echocardiography at week 52 as compared to baseline | at week 52
Change in aortic stenosis severity as measured by dimensionless velocity using echocardiography at week 104 as compared to baseline | at week 104 as compared to baseline
Change in coronary artery and mitral annulus calcium score at week 52 as compared to baseline | at week 52 as compared to baseline
Change in coronary artery and mitral annulus calcium score at week 104 as compared to baseline | at week 104 as compared to baseline
Change in serum DPP-4 at week 104 compared to baseline | at week 104 as compared to baseline
Change in serum IGF-1 at week 104 compared to baseline | at week 104 as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jae K Oh, MD, Principal Investigator — Mayo Clinic
Locations (25):
- United States (24):
  - Mayo Clinic, AZ, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, FL, Jacksonville, Florida
  - Baycare Health systems, Safety Harbor, Florida
  - Northside Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Rutgers- Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Ichan School of Medicine, New York, New York
  - Stony brook, Stony Brook, New York
  - Christ Hospital, Cincinnati, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Mechanicsburg, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Texas Heart Institute, Houston, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Inova Health Care Services, Falls Church, Virginia
  - Aurora Research Institute, Milwaukee, Wisconsin
- Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval, Québec, Canada